CLINICAL TRIAL: NCT01034956
Title: Outcomes and Patient Experience After Soft Tissue Dermal Filler Injections
Status: Completed | Type: Observational
Sponsor: The New York Eye & Ear Infirmary (Other)
Collaborators: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Anthony P. Sclafani, Director of Facial Plastic Surgery, The New York Eye & Ear Infirmary
Other Study IDs: 09.27
Record Dates: First submitted 2009-11-24; First posted 2009-12-18 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-04

CONDITIONS: Rhytids; Wrinkles
Keywords: Soft tissue filler; Dermal filler; Complications; Patient satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Facial Soft Tissue Filler Patients: Patients previously treated by Principal Investigator with facial soft tissue fillers within the past 2 years
  Interventions: Device: hyaluronic acid or calcium hydroxylapatite filler

INTERVENTIONS:
Device: hyaluronic acid or calcium hydroxylapatite filler — Intradermal and subdermal injection of facial soft tissue filler within the past 24 months; survey of patients to assess satisfaction and determine the presence of treatment related adverse events.
  Other Names: Restylane; Perlane; Juvederm; Radiesse

SUMMARY:
Purpose of the study:

The overall goal of this study is to better understand patient experience with injectable facial fillers so that the investigators may provide the best results for their patients. To do this, the investigators are administering surveys to approximately 50 patients who have been treated by Dr. Anthony P Sclafani, MD, FACS.

Participation:

Participants will be asked to complete a brief questionnaire regarding their most recent treatment by Dr. Sclafani with a facial injectable filler. All responses will be analyzed anonymously.

DETAILED DESCRIPTION:
Patients previously treated by the PI with dermal fillers will be mailed questionnaires about their experience with the treatment. These questionnaires will be deidentified prior to recording answers on a computer based spreadsheet.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated by Principal Investigator with facial soft tissue filler within the past 2 years willing to complete the research survey.

Exclusion Criteria:

* Any patient not treated by Principal Investigator with facial soft tissue filler within the past 2 years.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated by Principal Investigator with facial soft tissue filler within the past 2 years
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-11; Primary Completion 2010-03 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Satisfaction with treatment with facial soft tissue fillers | 0-24 months

SECONDARY OUTCOMES:
Social and behavioral effects of facial soft tissue filler treatment | 0-24 months

CONTACTS AND LOCATIONS:
Overall Officials: Anthony P Sclafani, MD, Principal Investigator — The New York Eye & Ear Infirmary
Locations (1):
- The New York Eye & Ear Infirmary, New York, New York, United States